CLINICAL TRIAL: NCT04568096
Title: Combination of Chemopreventive Agents (All- Trans Retinoic Acid and Tamoxifen) as Potential Treatment for the Lung Complication of COVID-19
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Kafrelsheikh University (Other)
Responsible Party: Principal Investigator, Mahmoud Ramadan mohamed Elkazzaz, Faculty of Science, Damietta University, Kafrelsheikh University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: COVID-2019
Record Dates: First submitted 2020-09-26; First posted 2020-09-29 (Actual); Last update posted 2020-10-26 (Actual); Status verified 2020-10

CONDITIONS: the Lung Complication of COVID-19
MeSH Terms: interventions — Tamoxifen

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Aerosolized All-Trans Retinoic acid plus oral Tamoxifen (Active Comparator): The infected patients will receive Aerosolized All-Trans Retinoic Acid in gradual in 2 divided doses increases from 0.2 mg/kg/day to 4 mg/kg/day as inhaled All-Trans Retinoic Acid therapy plus tamoxifen 20mg orally once daily. for 14 days
  Interventions: Combination Product: Aerosolized All-Trans Retinoic acid plus oral Tamoxifen
- The standard therapy (Placebo Comparator): The infected patients will receive the standard therapy for COVID-19 for 14 days
  Interventions: Other: Standard treatment

INTERVENTIONS:
Combination Product: Aerosolized All-Trans Retinoic acid plus oral Tamoxifen — After randomization and standard treatment The infected patients will receive Aerosolized All-Trans Retinoic Acid in gradual in 2 divided doses increases from 0.2 mg/kg/day to 4 mg/kg/day as inhaled All-Trans Retinoic Acid therapy plus tamoxifen 20mg orally once daily. for 14 days
  Arms: Aerosolized All-Trans Retinoic acid plus oral Tamoxifen
Other: Standard treatment — Standard treatment is according to the protocol of treatment of 2019-nCoV infection
  Arms: The standard therapy

SUMMARY:
Combination of Chemopreventive agents (All- Trans Retinoic Acid and Tamoxifen) as potential treatment for the Lung Complication of COVID-19

Abstract

Angiotensin-converting enzyme (ACE2) protein found on the cell membranes is the target of SARS-CoV-2 for entering into the host cells. Viral spike protein-binding with ACE2 down-regulates it. As ACE2 is known to protect the lung from injuries, SARS-CoV-2-induced ACE2 deficiency may expose patients to lung damage. In this Review, we use established and emerging evidence based on the findings of previous studies and researches to propose a testable hypothesis that Combination of chemopreventive agents (All Trans Retinoic acid and Tamoxifen) can be tested to prevent inflammatory complication in severe acute respiratory syndrome coronavirus 2 infection via two mechanisms by inhibiting bradykinin B1,B2 receptors expression and upregulating the depleted ACE2 in COVID-19 . Bradykinin B1 receptors are not expressed under physiological conditions but are induced under inflammatory conditions. Here we hypothesize that permanent attack and invasion of COVID-19 to lung epithelial cells via binding to ACE2 leads to tissue injury and inflammation and that increases BK levels and BK-B2-receptor (B2R) stimulation A study reported that tissue injury and inflammation increases BK levels and BK-B2-receptor (B2R) stimulation. We suggest that Bradykinin mediates and induces lung injury, proinflammatory cytokines and inflammation likely precipitates life threatening respiratory complications in COVID-19. Further experiments showed that BK treatment stimulated IL-6 production On the other hand a study reported that cells treated with Retinoic acid and Tamoxifen for 48 h significantly decreased the BK-B2 receptor protein levels (70.3 ± 0.6% vs. 100% of control, P < 0.05). Retinoids inhibit bradykinin B1 receptor-sensitized responses and this action could participate in their anti-inflammatory and immunomodulatory effects. In addition retinoic acid, is known to possess in vivo anti-inflammatory, anti-platelet and fibrinolytic activities. A study investigated the in vitro thrombin and platelet aggregation inhibitory activities of retinoic acid and retinaldehyde.Retinoic acid, retinaldehyde and retinol exhibited potent inhibition of thrombin, with IC50 values of 67μg/ml, 74μg/ml and 152μg/ml, respectively for the inhibition of thrombin (Sigma); and 49μg/ml, 74μg/ml and 178μg/ml, respectively for the inhibition of thrombin (plasma). Amongst vitamin A and its derivatives, retinoic acid showed the highest inhibition of both the forms of thrombin. Beside the effectiveness of TAM on cancer cells, it also has other effects on numerous microbes including parasite, fungi, bacteria, and some viruses such as Ebola virus and human immunodeficiency virus (HIV).Furthermore Tamoxifen can block the action of interleukin 6 and inhibit neutrophils. A study demonstrated that tamoxifen has side effects associated with neutropenia. Since tamoxifen can cause neutropenia and subsequently influence the neutrophil-to-lymphocyte ratio (NLR) value In addition it has anti malarial effect similar to chloroquine In conclusion

Keywords: COVID 2019 , Retinoic acid, Endosomal toll-like receptor 3,T Cells, IFN type1, AT1, ACE2,TMPRSS2

DETAILED DESCRIPTION:
This is a Phase 2, , randomized (1:1), placebo-controlled, 2-weeks, proof-of-concept study to evaluate the safety and tolerability as well as the mechanistic effect of Aerosol administration of Inhaled All trans retinoic acid and oral Tamoxifen in subjects infected with COVID -19

After randomization and standard treatment The infected patients will receive Aerosolized All-Trans Retinoic Acid in gradual in 2 divided doses increases from 0.2 mg/kg/day to 4 mg/kg/day as inhaled All-Trans Retinoic Acid therapy plus tamoxifen 20mg orally once daily. for 14 days

Inclusion Criteria:

Adult SARI patients with 2019-ncov infection confirmed by PCR; Absolute value of lymphocytes < 0. 6x 109/L; Severe respiratory failure within 48 hours and requires admission to ICU. (severe respiratory failure was defined as PaO2/FiO2 < 200 mmHg and was supported by positive pressure mechanical ventilation (including non-invasive and invasive mechanical ventilation, PEEP>=5cmH2O))

Exclusion Criteria:

Age < 18 Pregnant Allergic to experimental drugs and patients have the following conditions:

Hypercholesterolemia Hypertriglyceridemia Liver disease Renal disease Sjögren syndrome Pregnancy Lactation Depressive disorder Body mass index less than 18 points or higher than 25 points Contraindications for hormonal contraception or intrauterine device. Autoimmune diseases A history of organ, bone marrow or hematopoietic stem cell transplantation Patients receiving anti-hcv treatment Permanent blindness in one eye History of iritis, endophthalmitis, scleral inflammation or retinitis 15-90 days of retinal detachment or eye surgery The competent physician considered it inappropriate to participate in the study Previous history of deep vein thrombosis or pulmonary embolism in the last 12 months.

Patients with postmenopausal vaginal bleeding with no defined etiology. Patients with breast cancer who need to use tamoxifen for this neoplasm Another synchronous neoplasm that requires systemic treatment Patients with aggressive disease requiring cytotoxic therapy or locoregional therapies (eg hepatic embolization) A history of serious clinical or psychiatric illness that, by clinical judgment, may involve participation risk in this study Patients participating in other protocols with experimental drugs. Patients with oral food difficulties. Patients who underwent major recent surgery less than 4 weeks previously. Patients receiving chemotherapy or other oncologic therapy for less than 3 weeks

Study Type: Interventional Primary Purpose: Treatment Study Phase: Phase 2 Interventional Study Model: Parallel Assignment Number of Arms: 2 Masking: None (Open Label) Allocation: Randomized Enrollment: 160 [Anticipated]

ELIGIBILITY:
Inclusion Criteria:

Adult SARI patients with 2019-ncov infection confirmed by PCR; Absolute value of lymphocytes < 0. 6x 109/L; Severe respiratory failure within 48 hours and requires admission to ICU. (severe respiratory failure was defined as PaO2/FiO2 < 200 mmHg and was supported by positive pressure mechanical ventilation (including non-invasive and invasive mechanical ventilation, PEEP>=5cmH2O))

Exclusion Criteria:

Age < 18 Pregnant Allergic to experimental drugs and patients have the following conditions:

* Hypercholesterolemia
* Hypertriglyceridemia
* Liver disease
* Renal disease
* Sjögren syndrome
* Pregnancy
* Lactation
* Depressive disorder
* Body mass index less than 18 points or higher than 25 points
* Contraindications for hormonal contraception or intrauterine device.
* Autoimmune diseases A history of organ, bone marrow or hematopoietic stem cell transplantation
* Patients receiving anti-hcv treatment
* Permanent blindness in one eye
* History of iritis, endophthalmitis, scleral inflammation or retinitis 15-90 days of retinal detachment or eye surgery
* The competent physician considered it inappropriate to participate in the study Previous history of deep vein thrombosis or pulmonary embolism in the last 12 months.
* Patients with postmenopausal vaginal bleeding with no defined etiology.
* Patients with breast cancer who need to use tamoxifen for this neoplasm
* Another synchronous neoplasm that requires systemic treatment Patients with aggressive disease requiring cytotoxic therapy or locoregional therapies (eg hepatic embolization) A history of serious clinical or psychiatric illness that, by clinical judgment, may involve participation risk in this study
* Patients participating in other protocols with experimental drugs.
* Patients with oral food difficulties.
* Patients who underwent major recent surgery less than 4 weeks previously.
* Patients receiving chemotherapy or other oncologic therapy for less than 3 weeks

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Estimated)
Dates: Start 2020-11 (Estimated); Primary Completion 2020-12 (Estimated); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
lung injury score | at 7and 14 days
  Proportion of lung injury score decreased or increased after treatment

SECONDARY OUTCOMES:
Angiotensin 1-7 (Ang 1-7) changes over time | at day 7 and 14
Angiotensin 1-5 (Ang 1-5) changes over time | at day 7 and 14
Renin changes over time | at day 7 and 14]
Aldosterone changes over time | at day 7 and 14
Angiotensin-converting enzyme (ACE) changes over time | at day 7 and 14
Frequency of adverse events and severe adverse events | 14 days
Angiotensin II (Ang II) changes over time | at day 7 and 14
Sequential organ failure assessment score(SOFA score) over time | at day 7 and 14
Transe membrane protease ,serine II (TMPRSS2) changes over time | at day 7 and 14
Testosterone levels changes over time | day 7 and 14
Dihydrotestosterone(DHT) levels changes over time | day 7 and 14
Thrombin time (TT) | day 7 and 14

CONTACTS AND LOCATIONS:
Overall Officials: Mahmoud Elkazzaz, B.Sc in Biochemistry, Principal Investigator — Facculty of Science, Damietta University